CLINICAL TRIAL: NCT05157789
Title: The Effect of Informing Relatives of Patients With Short Messages on Anxiety Level During Cardiovascular Surgery
Brief Title: The Effect of Informing Relatives of Patients With Short Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Figen Dıgın, Assistant Professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KMarcinkowskiUMS
Record Dates: First submitted 2021-10-18; First posted 2021-12-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Surgery; Anxiety; Short Message
Keywords: Cardiovascular surgery; anxiety; relatives of the patient; Short message
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sms group (Experimental): Relatives of patients who were sent SMS
  Interventions: Other: SMS
- Control Group (No Intervention): Relatives of patients who were no intervation

INTERVENTIONS:
Other: SMS — In the study, text message will be sent to relatives of the patients for informing and the effect will be determine on the level of anxiety during cardiovascular surgery.
  Arms: Sms group

SUMMARY:
Surgical intervention is a planned or unplanned procedure performed to eliminate the existing or subsequent abnormal conditions in the individual's body, to reduce the effects of these conditions, or to remove the abnormal structures from the individual's body to eliminate the existing distress. While surgical interventions also cause anxiety in patients, it is known that they also cause significant anxiety in patients' relatives.This study was planned as a randomized controlled experimental study in order to examine the effect of this information on the anxiety level of the relatives of the patients by informing the relatives of the patients about the operation process with a short message during cardiovascular surgery.

In data collection; Introductory information form for the patient and patient relatives, a short message follow-up form, state and trait anxiety inventory will be used during the surgical intervention.

The sample of the study will be the relatives of the patients who are willing to participate in the study. Considering the change in the state anxiety scale scores between the experimental and control groups in the study of Baydemir S. (2019), it is calculated that there is a large effect size difference. Based on this finding, in order to test a large effect size (d=0.8) difference in anxiety scale scores of patient relatives between our experimental and control groups with 5% margin of error and 95% power, a total of 84 relatives of patients, 42 from each group, were included in the study. needed was calculated.

H0: Informing by text message has no effect on the anxiety of patient relatives.

H1: Informing by text message has an effect on the anxiety of patient relatives.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* To know Turkish,
* Being literate
* Having mental adequacy,
* Willingness to participate in the research,
* Having an active mobile line,
* Ability to use a telephone
* Being in the hospital before, during and after the operation

Exclusion Criteria:

* Be under the age of 18,
* Not knowing Turkish,
* Being illiterate
* Lack of mental adequacy,
* Lack of active mobile line,
* Inability to use the phone
* Absence from the hospital before, during and after the operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Anxiety of relatives of patients in the field of cardiovascular surgery assessed by the State Anxiety Inventory (SAI) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sisman C, Digin F. The Effect of Informing Patient Relatives with a Short Message on Anxiety Levels during Cardiovascular Surgery in Turkiye: A Randomized Controlled Trial. Niger J Clin Pract. 2024 Jun 1;27(6):708-715. doi: 10.4103/njcp.njcp_607_23. Epub 2024 Jun 29. PMID 38943294